CLINICAL TRIAL: NCT05801172
Title: Relieving Outpatient Hysteroscopy-associated Pain: What is the Most Effective Method?
Brief Title: Managing Outpatient Hysteroscopy-associated Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Jagiellonian University (Other)
Responsible Party: Principal Investigator, Iwona Magdalena Gawron, Ph.D., Principal Investigator, Jagiellonian University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1072.6120.228.2021
Record Dates: First submitted 2023-03-11; First posted 2023-04-06 (Actual); Last update posted 2023-08-08 (Actual); Status verified 2023-08

CONDITIONS: Pain; Hysteroscopic Surgery
MeSH Terms: conditions — Pain | interventions — Ketoprofen; Analgesia; Anesthesia, Local; Lidocaine; Anesthesia, Obstetrical

STUDY DESIGN:
Intervention Model Description: Women are randomly assigned to 3 arms - A: NSAID (ketoprofen 100 mg intravenously), B: A+infiltration anesthesia (20 ml 1% lidocaine), C: A+paracervical block (20 ml 1% lidocaine).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- A (NSAID) (Active Comparator): ketoprofen 100 mg intravenously 30 min. pre-office hysteroscopy
  Interventions: Procedure: ketoprofen plus infiltration anesthesia with lidocaine for pain relief in office hysteroscopy; Procedure: ketoprofen plus paracervical block anesthesia with lidocaine for pain relief in office hysteroscopy
- B (A+infiltration anesthesia) (Active Comparator): ketoprofen 100 mg intravenously 30 min. pre-office hysteroscopy plus 20 ml 1% lidocaine in intracervical administration at the start of the procedure
  Interventions: Procedure: ketoprofen for pain relief in office hysteroscopy; Procedure: ketoprofen plus paracervical block anesthesia with lidocaine for pain relief in office hysteroscopy
- C (A+paracervical block) (Active Comparator): ketoprofen 100 mg intravenously 30 min. pre-office hysteroscopy 20 ml 1% lidocaine in pericervical administration at the start of the procedure
  Interventions: Procedure: ketoprofen for pain relief in office hysteroscopy; Procedure: ketoprofen plus infiltration anesthesia with lidocaine for pain relief in office hysteroscopy

INTERVENTIONS:
Procedure: ketoprofen for pain relief in office hysteroscopy — ketoprofen ketoprofen 100 mg intravenously 30 minutes pre-procedure for pain relief in office hysteroscopy
  Arms: B (A+infiltration anesthesia); C (A+paracervical block)
Procedure: ketoprofen plus infiltration anesthesia with lidocaine for pain relief in office hysteroscopy — ketoprofen ketoprofen 100 mg intravenously 30 minutes pre-procedure for pain relief in office hysteroscopy plus 20 ml 1% lidocaine in intracervical administration at the start of the procedure
  Arms: A (NSAID); C (A+paracervical block)
Procedure: ketoprofen plus paracervical block anesthesia with lidocaine for pain relief in office hysteroscopy — ketoprofen ketoprofen 100 mg intravenously 30 minutes pre-procedure for pain relief in office hysteroscopy plus 20 ml 1% lidocaine in paracervical block at the start of the procedure
  Arms: A (NSAID); B (A+infiltration anesthesia)

SUMMARY:
Hysteroscopy is a reference diagnostic and therapeutic procedure in intrauterine pathologies, increasingly performed without general anesthesia. Pain is the most common reason for discontinuation of outpatient hysteroscopy (OH). There is no consensus on pain alleviation during OH. The aim was to compare the effectiveness of pain relief options during OH.

DETAILED DESCRIPTION:
A prospective randomized trial (consent no.1072.6120.228.2021) includes women subjected to OH due to focal uterine lesion, abnormal uterine bleeding, or infertility. Women are randomly assigned to 3 arms - A: NSAID (ketoprofen 100 mg intravenously), B: A+infiltration anesthesia (20 ml 1% lidocaine), C: A+paracervical block (20 ml 1% lidocaine). Karl Storz 5.0 mm Bettocchi® operative sheath with 2.9 mm 30 degree telescope and 5 Fr working channel was used. Intensity of pain in numeric rating scale (NRS), intensity of cervical bleeding, frequency of vaso-vagal reaction, and frequency of abandoning/ limiting the procedure were compared.

ELIGIBILITY:
Inclusion Criteria:

* age over 18
* indications for hysteroscopy: focal uterine lesion, abnormal uterine bleeding, or infertility

Exclusion Criteria:

* allergies to medications
* refusal to consent to the procedure or participation in the study

Ages: 18 Years to 90 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 201 (Actual)
Dates: Start 2022-07-01 (Actual); Primary Completion 2023-06-01 (Actual); Study Completion 2023-07-01 (Actual)

PRIMARY OUTCOMES:
Intensification of pain in Numeric Rating Scale: 0-10 | up to 6 months
  Measurement and comparison of the intensity of pain in numeric rating scale (NRS) during and after the procedure in 3 study arms

SECONDARY OUTCOMES:
Intensity of cervical bleeding on the assumed scale: 0-3 | up to 6 months
  Measurement and comparison of the intensity of cervical bleeding (intensity scale: 0-3) during the procedure in 3 study arms
Occurrence of vaso-vagal reaction during the procedure | up to 6 months
  Measurement and comparison of the frequency of vaso-vagal reaction during the procedure in 3 study arms
Occurrence of abandoning/ limiting the procedure | up to 6 months
  Measurement and comparison of the frequency of abandoning/ limiting the procedure due to pain in 3 study arms

CONTACTS AND LOCATIONS:
Overall Officials: Robert Jach, Prof., Study Chair — Jagiellonian University
Locations (1):
- Jagiellonian University Medical College, Department of Gynecology and Obstetrics, Krakow, Poland

IPD SHARING:
Plan to Share IPD: No